CLINICAL TRIAL: NCT02081716
Title: Assessment of CMV-specific ELISPOT Assay for Predicting CMV Infection in Bone Marrow Transplant Recipients (ACE-BMT)
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Han Kim, Assocaite Professor, Asan Medical Center
Other Study IDs: 2014-0103
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Bone Marrow Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- high CMV ELISPOT results: high spot counts in ELISPOT
- low CMV ELISPOT results: low spot counts in ELISPOT

SUMMARY:
CMV is one of the most important opportunistic infection in transplant recipients. In South Korea, more than 95% of adults reveal sero-positivity for CMV IgG. Until now, sero-positivity for CMV IgG before bone marrow organ transplantation is a laboratory test of choice to stratify the risk of CMV reactivation after solid organ transplantation. Theoretically, CMV-specific cell-mediate immune response before and after bone marrow transplantation will further categorize the patients into high or low risk of CMV development after bone marrow transplantation. The investigators thus evaluate the usefulness of CMV-specific ELISPOT assay in bone marrow transplant candidates to predict the development of CMV infection after transplantation.

DETAILED DESCRIPTION:
We will evaluate whether CMV-specific cell-mediated immune response before transplant, 1 month, 3 months, and 6 months after transplantation will predict CMV infection after bone marrow transplantation.

ELIGIBILITY:
Inclusion Criteria:

* age 16 or more
* agree with written informed consent

Exclusion Criteria:

* no exclusion criteria

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: bone marrow transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
CMV infection | 6 months after transplantation
  CMV infection is defined as follows.
  1. CMV viremia: CMV antigenemia or CMV quantitative PCR (+)
  2. CMV disease: CMV syndrome or tissue-invasive CMV disease i) CMV syndrome: ① CMV viremia ② temperature > 38 without other cause ③ WBC < 4000, atypical lymphocyte > 3%, transaminase elevation, platelet < 100,000/mm ii) tissue-invasive CMV disease: evidence of CMV in histopathologic specimen (inclusion body or viral antigen in biopsy or bronchoalveolar lavage fluid)

SECONDARY OUTCOMES:
mortality | 6 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Han Kim, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea